CLINICAL TRIAL: NCT06263647
Title: Launching the Houston-HVIP: Developing and Evaluating a Hospital-Based Intervention to Reduce Recurrent Violence
Brief Title: Launching the Houston Hospital-Based Violence Intervention Program (Houston-HVIP): Developing and Evaluating a Hospital-Based Intervention to Reduce Recurrent Violence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Sandra L. McKay, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HSC-MS-23-0904; UG3NR021232 (NIH); UH3NR021232 (NIH)
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-05

CONDITIONS: Firearm Injury
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be partially blinded in that they will know some information about the intervention but will not be exposed to the details of the intervention or the intervention manual.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Houston-HVIP treatment group (Experimental)
  Interventions: Behavioral: Houston-HVIP treatment
- Standard of Care group (Active Comparator)
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Houston-HVIP treatment — Participants will be assigned a case manager to provide a brief assessment of , psychological and social needs and a risk assessment and create individualized discharge planning. Participants will be referred to tailored social service programs based on the needs, including assessments of social determinants of health, educational and financial needs, and subsequent referral for programs such as job training, educational support, housing assistance, or financial assistance programs for identified needs. Participants identified at risk for violence perpetration via a risk assessment screener will be referred to the violence interrupter services. Long-term opportunities for engagement with the trauma survivors' network within Memorial Hermann Hospital will be available and encouraged.Participants will receive a structured curriculum that will include regular check-in with an assigned case manager over 6 months to promote successful community-based program integration and completion.
  Arms: Houston-HVIP treatment group
Behavioral: Standard of Care — Participants will be assigned a case manager to meet with the injured patients to briefly assess (a) psychological and social needs and (b) a risk assessment and create individualized discharge planning. Resources for the patient to connect with social service programs will be provided by the case manager. Long-term opportunities for engagement with the trauma survivors' network within Memorial Hermann Hospital will be available and encouraged. Follow-up contacts and services from an assigned case manager over two weeks following discharge from the hospital to ensure that the patient has contacted the community-level violence outreach organizations.
  Arms: Standard of Care group

SUMMARY:
A prior violent injury is one of the strongest predictors of future violent injury, highlighting the importance of effective hospital-based interventions to prevent reinjury. This project will establish and evaluate the Houston Hospital-Based Violence Intervention Program (Houston-HVIP). Using a randomized controlled trial, the study will assess the effectiveness of Houston-HVIP in reducing violent reinjury and improving behavioral, mental, and physical health outcomes over a 12-month follow-up period among those enrolled in the study in ages 16-35 years of age.

ELIGIBILITY:
Inclusion Criteria:

* presented for a gunshot injury stemming from community violence at Memorial Hermann Hospital
* English or Spanish-speaking
* provide informed voluntary consent to participate in the study
* live in Harris County at time of enrollment

Exclusion Criteria:

* presenting for a firearm injury arising from a self-inflicted gunshot or unintentional gun violence
* actively detained by criminal justice systems at time of enrollment

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 274 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in repeat violent victimization as assessed by the number of participants who return to the hospital system for for an intentional firearm injury | Baseline , 3 months, 6 months, 9 months and 12 months

SECONDARY OUTCOMES:
Change in repeat non-firearm violent victimization as assessed by the number of participants who return to the hospital system for an intentional non-firearm injury | Baseline , 3 months, 6 months, 9 months and 12 months
Change in attitudes towards firearm violence as assessed by Firearm Violences Attitudes (Sheley; Shapiro) questionnaire | Baseline , 3 months, 6 months, 9 months and 12 months
  This is a 13-item questionnaire; however, only items 3,4,7,9,10,12 and 13 will be asked. Each is scored from 1(strongly disagree) - 4(strongly agree), Maximum score of 28 .Higher score indicates more aggression.
Change in post-traumatic stress as assessed by the post-Traumatic Stress Disorder Checklist Version 5(PCL-5) | Baseline , 3 months, 6 months, 9 months and 12 months
  This is a 20-item questionnaire; however only items 1 and 4 of the PCL-20 will be asked. These 2 items will be anchored to a stressful experience. And each is scored form 0(not at all)-4(extremely), maximum score of 8, higher score indicating worse outcome
Change in aggression as assessed by the Copeland-Linder questionnaire. | Baseline , 3 months, 6 months, 9 months and 12 months
  This is a 7-item questionnaire; however, only items 1, 5, and 6 will be asked. Each is scored from 1(strongly disagree) - 4(strongly agree). Maximum score is 12. Higher score indicates more aggression
Change in general health as assessed by the 12-item Short Form Health Survey (SF-12) | Baseline , 3 months, 6 months, 9 months and 12 months
  This is a 12 item questionnaire; however, only item #1 will be asked. It is scored from 1(excellent) - 5(poor), higher number indicating worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Sandra McKay, MD, Principal Investigator — The University of Texas Health Science Center, Houston; Alexander Testa, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No